# **Document Date: 05/12/2023** 1 2 Investigation of the Effect of Radial Nerve Mobilization on Pain, Function, and Grip Strength in Patients with Thumb Osteoarthritis: A Randomized Controlled Trial 3 4 Ethics Approval: The study was conducted with the approval of the Ethics Review Board of 5 Gazi University, Ankara, Turkey. (approval number 2022 - 1117). 6 Clinical trials ID: NCT05650970 7 8 MATERIALS AND METHODS 9 10 The design of this prospective, randomized controlled, single-blinded parallel study was approved by the Gazi University Ethics Committee (Date: 04.10.2022, Research Code No: 11 2022 - 1117). 12 This study was conducted with patients who applied to the Hand Surgery Outpatient Clinic of 13 X hospital between November 2022 and February 2023 and were referred to hand therapy 14 15 with the diagnosis of TMC OA in Ankara. The patients included in the study were divided into two groups: mobilization and control groups according to the order in which they applied 16 17 to the clinic. The treatment and evaluation of all patients were carried out by two different hand therapists 18 at X University Hand Rehabilitation Unit. The evaluations were made twice, before treatment 19 and after four weeks of the treatment. The patients in both groups received treatment 2 20

sessions per week for 4 weeks. All patients were called for a second evaluation on a separate

day after the completion of their treatment to avoid an acute effect of the treatment session on

21

22

23

the results.

### **Participants**

26 The inclusion criteria of the participants were the diagnosis of OA in the TMC joint and the presence of pain. It was planned to exclude patients who had a history of surgery (trigger 27 finger, carpal tunnel, Dupuytren's contracture, tenosynovitis, etc.) in the last 6 months, using 28 a splint for thumb during the previous 3 months, and who had lack of cooperation, which 29 could be an obstacle to completing the questionnaires. In addition, patients who were found to 30 have any extra pathologies of the upper extremity (epicondylitis, neck hernia, nerve 31 32 compression, bone cyst, etc.) that could cause pain during the study period and who started to use splinting, pain relieving treatments such as medications or injection were excluded from 33 the study. Evaluation and treatment of patients with bilateral involvement were done for both 34 hands and each hand's results were recorded separately. Among the data of these patients, 35 clinical status (symptomatic hand, stage, and symptom duration), pain (at rest, activity, and 36 37 night), strength (gross grip, lateral, and double pinch), and performance in the Nine-Hole Peg 38 Test (9HPT) were included in the analysis for both hands separately; demographic information (age, height, weight, gender) and scores of Michigan Hand Outcomes 39 Questionnaires (MHOQ) and Functional Index of Hand Osteoarthritis (FIHOA) were included 40 as single data for each patient. 41 The entire flow data of the patient enrollment is given in Figure 3 as a flowchart according to 42 the CONSORT guide. 43 The patients were informed about the study on the first day they came to the hand 44 45 rehabilitation unit for treatment, and their written consent was obtained. The patient's age, gender, height, body weight, dominant and affected hand, surgical history, previous 46

treatments, disease stage, and duration of symptoms were recorded. Afterward, physical
 assessments were performed.

49

50

#### **Outcome measures**

In this study, our primary outcome measure was the improvement in pain level; secondary 51 52 outcome measures were the improvement in thumb function and grip strength. The pain level of the participants was evaluated with the Visual Analog Scale (VAS) in 3 53 different conditions including rest, activity, and night. The assessment was made with a 10-cm 54 straight line with endpoints describing the intensity of the pain. All patients were asked to mark 55 the pain level corresponding to the intensity of the pain on the line between "0" representing 56 "no pain" and "10" representing "the most/extremely unbearable pain". The distance between 57 "0" and the mark made by the patients was measured and recorded in cm. 58 A hydraulic hand dynamometer (Jamar ®) was used for grip strength assessment, and a pinch 59 meter was used for bipod and lateral pinch strength. These measurements were made in the 60 standard sitting position as determined by the American Association of Hand Therapists. The 61 participant holds the elbow at 90 degrees flexion and the wrist in a neutral position at the side 62 of the trunk. During the assessment, the patient sits in a chair with a backrest. During the grip 63 strength measurements, the patient was asked to squeeze as hard as possible, and the 64 65 measurements were repeated three times consecutively for both hands. The mean value of the measurement results was taken and recorded in kilograms (kg). 66 9HPT was used in the evaluation of the functionality and fine dexterity level of each hand. 67 During this evaluation, the patient sits in a comfortable position. The patient was taught the 68 test to be performed and allowed to make a trial. Starting from the position where the pegs 69 were inserted into the holes, the patient was asked to remove all the pegs as fast as he/she 70

could with the evaluated hand, remove the last one, and then quickly insert the pegs into the

holes. The total removal and insertion times were recorded in seconds for both hands

73 separately.

72

74

75

76

77

78

79

80

81

82

83

84

85

86

87

88

89

90

91

92

93

The FIHOA questionnaire developed specifically for hand osteoarthritis was used to assess

the level of disability. The questionnaire consists of 10 items containing statements about the

use of hands in daily life, and each item is scored from 0 to 3 points according to the difficulty

level: "0: possible without difficulty", "1: possible with slight difficulty", "2: possible with

importance difficulty", "3: impossible". The total score varies from 0 to 30 points. As a result

of this questionnaire, a low score represents a better function, while a high score represents a

worse function. The adapted version of the Turkish language was used.

The Michigan Hand Outcomes Questionnaires (MHOQ) were used in the functionality and

general evaluation of hand use bilaterally and right-left separately in daily life. The MHOQ is

reliable, valid, and responsive in patients with TMC joint osteoarthritis. The questionnaire

evaluates pain, function, aesthetic appearance, and satisfaction as sub-parameters. Since the

MHOQ measures function/satisfaction, the higher the score on the questionnaire, the higher

the reported functionality/satisfaction. The adapted version to the Turkish language was used.

**Interventions** 

The study consisted of two groups: mobilization and control group. The only difference

between the mobilization group from the control group was the addition of radial nerve

mobilization exercises to the treatment program in this group. The remaining treatment

program was the same in both groups. Both groups in the study were included in the treatment

program twice per week for 4 weeks in the clinic. Patients were also instructed to repeat the

- exercises and interventions at home 3 times per day. The treatment program for the patients consists of the interventions below:
- Patient education: During the treatment period, patients were told not to use their hands for
  heavy work and not to perform any application other than the treatment. Patients were
  assessed about how much they use the hand during the day in daily life, during the recreation
  and hobby times and they were educated about the correct grip positions as explained below.
- Teaching correct grip techniques: Patients were taught correct gripping techniques with
   objects of different sizes and shapes and were informed about maintaining this position during
   their daily activities (Figures 1 and 2).
  - Massage: Massage was applied on the superficial branch of the radial nerve trace and the thumb. Relaxation in the tissue, pain relief with mechanical stimulation, and edema reduction were aimed.
    - Nerve mobilization exercise: Radial nerve mobilization exercises were performed in two consecutive ways: isolated wrist (ulnar-radial deviation with the thumb grasped in the palm in a fist) and combined wrist-elbow (wrist in ulnar deviation with the elbow in extension and wrist in radial deviation with the elbow in flexion, starting in anatomical posture). These exercises were only given to the mobilization group.
- Ice therapy: It was applied on the dermatome of the superficial branch of the radial nerve for
   10-12 minutes at the end of the treatment.

### Data analysis

SPSS 26.0 program was used for statistical analysis of the data. The measured data were expressed as percentages (%) and numbers (n) for qualitative variables and mean  $\pm$  standard

deviations for quantitative variables. The Pearson Chi-Square test was used for the comparison of the categorical variables (gender, dominant hand, affected hand, bilateral involvement, and history of surgery for the disease). All participants with available baseline data were included in the analyses. Missing outcomes were imputed based on baseline values. No participant was excluded from the final analysis because of missing data. The Mann-Whitney U test was used to compare the differences (delta) before and after the treatment. The magnitude of effect sizes of differences between groups was calculated using Monte Carlo defining clinically meaningful effect sizes with 95% Confidence level. P value <0.05 was accepted for statistical significance.

127 RESULTS

Sixty-four patients were invited to the study. A total of 6 patients were excluded because 2 of these patients did not meet the inclusion criteria (concomitant bone cyst in one patient and diagnosis of entrapment neuropathy in one patient) and 4 patients refused to participate in the study. After exclusion, 58 patients were included in the study. At the end of the 4-week treatment program, the data of 51 patients who completed the treatment program. Missing data of the 7 patients who discontinued were also included in the analysis after multiply imputation by maximum-likelihood-based regression methods. As a result, data from a total of 58 patients were analyzed. The remaining 58 patients were included in the mobilization (n=28) or control group (n=30). The patients did not know which group they belonged to. One patient in the mobilization group was excluded after the start of the study as she received an additional treatment. One another patient in this group discontinued the treatment program. Five patients in the control group discontinued the treatment. All participants with available baseline data were included in the analyses. Missing outcomes were imputed based on baseline values. No participant was excluded from the final analysis because of missing data.

Finally, the data of 58 patients in total, 28 in the mobilization group and 30 in the control 142 143 group were compared. Since 3 patients in the mobilization group and 1 patient in the control group had bilateral involvement, the evaluation and treatment of these patients were 144 performed separately for both hands. Therefore, the data from 58 patients (mobilization: 28, 145 control: 30) and 62 hands (mobilization: 31, control: 31 hands) were analyzed. (Figure 3). 146 Both groups were similar regarding their demographic and clinical characteristics (p>0.05). 147 148 The two groups differed only in the number of participants with a history of surgery for TMC OA. The number of patients who had surgery in the control group was 6 (20%) and 1 (3.57%) 149 in the mobilization group (p=0.045) (Table 1). Moreover, both groups were at similar clinical 150 151 levels in terms of the results of the pre-treatment evaluations in all parameters (p>0.05) (Table 2). 152 Comparison of the differences between the two groups before and after the treatment showed 153 that the improvement in pain level in rest (p=0.002), in activity (p=0.008), at night (p=0.053); 154 155 and gross grip (p=0.013) and lateral pinch strength (p=0.003); FIHOA score (p=0.001); and 156 MHOQ overall score (p=0.005) in the mobilization group were significantly superior to the control group (Table 3). 157

Figure 1: Gripping position before patient education

158



Figure 2: Gripping position after patient education



Figure 3: CONSORT flow-diagram of participants throughout the study period



Tablo 1: Baseline characteristics of the study groups

| Baseline characteristics | Mobilization group (n=28) | Control group (n=30) | P-<br>value | Z-<br>value | Effect size<br>[CI] |
|---|---|---|---|---|---|
| Age (years) (Mean ± SD) | 57.50 ± 11.30 | 61.67 ± 9.82 | 0.249 | -1.153 | 0.45<br>[0.44;0.46] |
| Height (cm) | 161.21 ± 9.41 | $160.83 \pm 8.26$ | 0.956 | -0.055 | 1[1] |
| Body weight (kg) | 73.64 ± 12.94 | 74.90 ± 8.14 | 0.586 | -0.545 | 0.40<br>[0.39;0.41] |
| Gender (n) (%)<br>(female/male) | 22/6 (78.5%) | 25/5 (83%) | 0.644 | | |
| Surgical history (n) (%) (operated/nonoperated) | 1/27 (3.57%) | 6/24 (20%) | 0.045* | | |
| Symptom duration (months) | 15.46 ± 13 | 15.93 ± 13.99 | 0.994 | -0.008 | 0.62<br>[0.61;063] |
| Dominant side (n) (%) | | | | | |
| Right | 26 (92.85%) | 29 (96.66%) | 0.513 | | |
| Left | 2 (7.15%) | 1 (3.34%) | | | |
| Symptomatic side (n) (%) | | | | | |
| Right | 14 (50%) | 12 (40%) | 0.305 | | |
| Left | 11 (39.28%) | 17 (56.66%) | | | |
| Bilateral | 3 (10.72%) | 1 (3.34%) | | | |
| Dominant hand<br>symptomatic (n) (%)<br>Yes | 16 (57.14%) | 13 (43.33%) | 0.201 | | |
| No | 9 (32.14%) | 16 (53.33%) | | | |
| Bilateral | 3 (10.72%) | 1 (3.34%) | | | |

| Grade (Eaton-Littler classification) (n) (%) | | | |
|---|---|---|---|
| Grade 1 | 1 (3.57%) | 3 (10%) | |
| Grade 2 | 8 (28.57%) | 14 (46.66%) | 0.288 |
| Grade 3 | 17 (60.72%) | 12 (40%) | |
| Grade 4 | 2 (7.14%) | 1 (3.34%) | |

n: Number of participants, SD: Standart Deviation, p<0.05: statistically significant, CI: Confidence Interval

# Table 2: Baseline values and between-group comparison results

| Baseline Values | Mobilization<br>group (n=31)<br>(Mean ± SD) | Control group<br>(n=31)<br>(Mean ± SD) | P value | Z value | Effect size [CI] |
|---|---|---|---|---|---|
| Pain in Resting (cm) | $3.34 \pm 2.33$ | $2.93 \pm 2.61$ | 0.373 | -0.891 | 0.37<br>[0.36;0.38] |

| Pain in Activity (cm) | $7.07 \pm 2.14$ | $6.70 \pm 1.85$ | 0.597 | -0.529 | 0.59<br>[0.58;0.60] |
|---|---|---|---|---|---|
| Pain in Night (cm) | $2.88 \pm 2.83$ | $2.74 \pm 3.23$ | 0.405 | -0.833 | 0.41<br>[0.40;0.41] |
| Grip Strength (kg) | $18.90 \pm 9.05$ | $19.85 \pm 7.52$ | 0.517 | -0.648 | 0.51<br>[0.51;0.53] |
| Bipod Pinch Strength (kg) | $3.16 \pm 1.29$ | $3.02 \pm 1.35$ | 0.582 | -0.550 | 0.58<br>[0.57;059] |
| Lateral Pinch Strength (kg) | $5.29 \pm 2.04$ | $5.40 \pm 1.86$ | 0.622 | -0.493 | 0.62<br>[0.61;0.63] |
| 9HPT Time (second) | $23.62 \pm 4.15$ | 24.33 ± 5.29 | 0.598 | -0.528 | 0.61<br>[0.60;0.62] |
| FIHOA Score | $13.39 \pm 6.06$ | $10.61 \pm 6.45$ | 0.057 | -1.906 | 0.055<br>[0.050;0.059] |
| MHOQ Overall Score | $49.37 \pm 13.20$ | 53.04 ± 10.40 | 0.145 | -1.457 | 0.14<br>[0.14;015] |

SD: Standart Deviation, MHOQ: Michigan Hand Outcomes Questionnaires, FIHOA: Functional Index of Hand Osteoarthritis, 9HPT: 9 Holes Peg Test, \*p<0.05: statistically significant, CI: Confidence Interval

Tablo 3: Result of comparing the differences between the pre- and post-treatment outcome

measures between the groups

| Outcome measures | Differences between Pre and post- treatment in mobilization group (Mean ± SD) | Differences<br>between Pre<br>and post-<br>treatment in<br>control group<br>(Mean ± SD) | P value | Z<br>value | Effect size |
|---|---|---|---|---|---|
| Pain (cm) | | | | | 0.002 |
| Resting | $1.89 \pm 2.10$ | $-0.02 \pm 2.43$ | 0.002* | -3.055 | [0.001;0.002] |
| Activity | $3.26 \pm 2.34$ | $1.64 \pm 1.87$ | 0.008* | -2.657 | [0.007;0.011] |
| Night | $2.19 \pm 2.43$ | $0.90 \pm 1.44$ | 0.053* | -1.935 | 0.055<br>[0.051;0.059] |
| Gross Grip Strength<br>(kg) | 4.31 ± 3.01 | $1.86 \pm 4.68$ | 0.013* | -2.487 | 0.009 [0.007;0.01] |
| Bipod Pinch Strength (kg) | $0.68 \pm 0.92$ | $0.22 \pm 1.33$ | 0.074 | -1.786 | 0.073 [0.068;0.078] |
| Lateral Pinch Strength (kg) | $1.29 \pm 1.65$ | $0.05 \pm 1.16$ | 0.003* | -2.954 | 0.002<br>[0.001;0.002] |
| 9HPT Time (second) | $2.52 \pm 3.35$ | $1.48 \pm 3.02$ | 0.192 | -1.303 | 0.198 [0.19;0.020] |
| FIHOA Score | $5.54 \pm 4.03$ | $2.06 \pm 4.20$ | 0.001* | -3.237 | 0.001 [0.001;0.002] |
| MHOQ Overall Score | $13.62 \pm 9.49$ | 5.91 ± 11.05 | 0.005* | -2.811 | 0.005 [0.003;0.006] |

n: Number of participants, SD: Standart Deviation, MHOQ: Michigan Hand Outcomes Questionnaires, FIHOA: Functional Index of Hand Osteoarthritis, 9HPT: 9 Holes Peg Test, \*p<0.05 statistically significant, CI: Confidence Interval